CLINICAL TRIAL: NCT06366555
Title: The Role of Manual Twirling Acupuncture in Reducing Biceps Brachii Muscle Pain and Stiffness After Weight Training in Healthy Untrained Individuals
Brief Title: The Role of Manual Twirling Acupuncture in Reducing Muscle Pain and Stiffness After Biceps Curling in Healthy Untrained Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Ray Sirvel, Doctor, Indonesia University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 24-02-0268
Record Dates: First submitted 2024-04-11; First posted 2024-04-16 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Muscle Soreness; Stiffness of Elbow, Not Elsewhere Classified
MeSH Terms: conditions — Myalgia

STUDY DESIGN:
Intervention Model Description: This research design used a randomized controlled single-blind crossover trial method (Crossover Single Blinded Randomized Control Trial). Reasons for choosing to use the Crossover method because apart from being able to implement it, it can also provide far more output results with a smaller number of subjects.
  The research subjects will then receive two treatments spaced 1 week apart which is called a wash out period to eliminate the carry-over effect of the treatment given. Research subjects will undergo randomization . Subjects in group A will undergo manual twisting acupuncture followed by sham manual acupuncture. The subject in group B will receive a sham acupuncture manual followed by a round of manual acupuncture twirling
Who Masked: Participant, Outcomes Assessor
Masking Description: The Participant will be randomized using a computerized table and the Outcome Assessor dont know which Subjects receive the manual acupuncture twirling or sham manual acupuncture on each period
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual acupuncture twirling (Experimental): In the intervention group, acupuncture needles were inserted using a tube with manipulation parameters, puncture is carried out using a sized needle 0.14 x 25 mm penetrates the plaster and skin with using the help of a 30 mm long tube to achieve a puncture depth of 20 mm and a twirling manipulation is carried out. For kinematic parameters of rotational movement in the same direction clockwise (to the right) by 180 degrees, 3 rad/s for 30 seconds at points PC2 and LU5.
  The time parameters were retained for 20 minutes and twirling was manipulated 0 minutes and 10 minutes. After the retention is over, control the bleeding with Press on the needle insertion point for 10 seconds or until the bleeding stops
  Interventions: Procedure: Manual Acupuncture Twirling,
- Manual acupuncture sham (Sham Comparator): in the sham group acupuncture needles were inserted using a tube without any manipulation parameters and not penetrating the skin. The needles then left for 20 minutes.
  Interventions: Procedure: Manual Acupuncture Sham

INTERVENTIONS:
Procedure: Manual Acupuncture Twirling, — Manual Acupuncture twirling : using 0.14x 25 mm needle, punctured and penetrated the skin and then a twirling manipulation is carried out, 180 degrees, 3 rad/second, for 30 second each at LU5 and PC2. The needles retained for 20 minutes and manipulated at 0 minutes and 10 minutes.
  Arms: Manual acupuncture twirling
Procedure: Manual Acupuncture Sham — Manual Acupuncture Sham : Using 0.14x25mm needles on plesterin without being penetrated into skin and no manipulation given, retained for 20 minutes
  Arms: Manual acupuncture sham

SUMMARY:
Regular physical activity can help to prevent and control non-communicable disease. WHO recommends at least in adults to do moderate-vigorous physical activity includes muscle strengthening. But regardless the importance and recommendations of physical activity, not all of the world's population does it .Biceps Curling is a popular physical exercise which easy to do , it can strengthen the muscles in the upper body. However based on the International Association for the Study of Pain (IASP) in individuals who just starting to do physical exercise may experience pain and can become a barrier to do physical activity, so an approach is needed to prevent this and acupuncture is one of them. Currently, a lot of acupuncture research has been carried out to reduce the condition pain and stiffness after weight training, but there are not many study using manual acupuncture twirling in this condition .

That's why the aim of this study Is to see the efficacy of giving manual acupuncture with twirling stimulation for pain and stiffness post weight training. The study method will be a Single Blinded Crossover Randomized Controlled Trial which will compare the efficacy of Manual Acupuncture twirling with Manual Acupuncture Sham for post-exercise pain and stiffness . The outcomes consist of Visual Analog Scale, Pain Pressure Threshold, Range of motion of elbow flexor at 24 hours, 48 hours, and 72 hours post weight training

DETAILED DESCRIPTION:
This is a clinical trial study with cross-over design with 1 week wash out period to evaluate and compare the effects of Manual Acupuncture twirling and Manual Acupuncture sham for pain and stiffness after Biceps Curling (Weight Training) on healthy untrained subjects. The subjects are 48 males/female and will be randomly assigned to 2 groups: (1) Manual Acupuncture Twirling/Manual Acupuncture Sham and (2) Manual Acupuncture Sham/Manual Acupuncture twirling group . The subjects will receive two times treatment on day 1 and day 7. The outcome will be assessed each before treatment (baseline) at 24 hours, 48 hours, and 72 hours post weight training. Patients and the outcome assessors will be blinded to the group allocation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Individuals with no exercise program
* Elligible for physical exercise
* Willing to take part in the study and sign informed consent

Exclusion Criteria:

* Consuming anti-inflammatory drugs, muscle relaxants and received any type of acupuncture within 7 days before the study
* Having contraindications of manual acupuncture (Pregnant, malignancy, bleeding disorders, needle phobia)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2024-04-22 (Actual); Primary Completion 2024-06-22 (Actual); Study Completion 2024-06-22 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | 0,24hours,48 hours, 72 hours
  Subjective Pain rated by score , Minimum Value 0, Maximum Value 10. 0 : No Pain, 10 : The Worst Pain Possible

SECONDARY OUTCOMES:
Pain Pressure Threshold | 0,24hours,48 hours, 72 hours
  Objective Pain

OTHER OUTCOMES:
Range of Motion | 0,24hours,48 hours, 72 hours
  Range of Elbow Flexor Extension

CONTACTS AND LOCATIONS:
Overall Officials: KEPK FKUI-RSCM, Principal Investigator — The Ethics Committee of the Faculty of Medicine, University of Indonesia - Cipto Mangunkusumo Hospital
Locations (1):
- Sport and Exercise Studies, Indonesian Medical Education and Research Institute (IMERI) Research Tower, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol